CLINICAL TRIAL: NCT03764735
Title: A Phase 3, Multi-Center, Randomized, Double-Masked, Placebo-Controlled Clinical Study to Assess the Safety and Efficacy of SkQ1 Ophthalmic Solution for the Treatment of Dry Eye Syndrome
Brief Title: Study of SkQ1 as Treatment for Dry-eye Syndrome
Acronym: VISTA-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mitotech, SA (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-110-0004
Record Dates: First submitted 2018-11-30; First posted 2018-12-05 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye; Dry Eye Syndrome; SkQ1; KCS; Keratoconjunctivitis
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis | interventions — Visomitin

STUDY DESIGN:
Intervention Model Description: Parallel-group study of two strengths of ophthalmic solution versus placebo solution
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SkQ1 Vehicle (Placebo Comparator): SkQ1 (Vehicle)
  Interventions: Drug: SkQ1 (Vehicle)
- Low Dose - SkQ1 (Active Comparator): Low-dose ophthalmic solution
  Interventions: Drug: Low Dose - SkQ1
- High Dose - SkQ1 (Active Comparator): High-dose ophthalmic solution
  Interventions: Drug: High dose - SkQ1

INTERVENTIONS:
Drug: Low Dose - SkQ1 — SkQ1 Low dose ophthalmic solution
  Other Names: Visomitin
  Arms: Low Dose - SkQ1
Drug: High dose - SkQ1 — SkQ1 High Dose ophthalmic solution
  Other Names: Visomitin
  Arms: High Dose - SkQ1
Drug: SkQ1 (Vehicle) — Vehicle for SkQ1 ophthalmic solution
  Arms: SkQ1 Vehicle

SUMMARY:
The purpose of this study is to evaluate whether SkQ1 ophthalmic solutions are safe and effective compared to placebo for the treatment of the signs and symptoms of dry eye syndrome.

DETAILED DESCRIPTION:
Multi-center, double-masked, randomized, placebo-controlled study comprising 5 visits over the course of approximately 9 weeks. Qualified subjects are randomized 1:1:1 to receive either High Dose SkQ1 ophthalmic solution, Low Dose SkQ1 ophthalmic solution, or Placebo (vehicle of SkQ1 ophthalmic solution).

The Primary Endpoints are:

Change from Baseline (Visit 2) to Visit 5 in Corneal Fluorescein Staining;

Change from Baseline (Visit 2) to Visit 5 in Grittiness Symptom

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent;
* Have a subject reported history of dry eye;
* Have a history of use of eye drops for dry eye symptoms ;
* Ocular Discomfort;
* Schirmer's Test score;
* Have corneal fluorescein staining ;
* Have lissamine green conjunctival Staining ;
* Have a conjunctival redness;

Exclusion Criteria:

* Have participated in the previous SkQ1 ophthalmic solution Phase 2 treatment study;
* Have any clinically significant slit lamp findings at Visit 1;
* Be diagnosed with an ongoing ocular infection or active ocular inflammation at Visit 1;
* Have had any ocular and/or lid surgeries within 6 months of Visit 1 or any planned over the study period;
* Have an uncontrolled systemic disease;
* Be a woman who is pregnant, nursing or planning a pregnancy;
* Be a woman of childbearing potential who is not using an acceptable means of birth control;
* Have a known allergy and/or sensitivity to the study drug or its components ;
* Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days of Visit 1;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-02-09 (Actual); Study Completion 2019-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence T Friedhoff, MD, PhD, Study Chair — Mitotech, SA
Locations (7):
- United States (7):
  - Cornea & Cataract Consultants of Arizona, Phoenix, Arizona
  - Eye Research Foundation, Newport Beach, California
  - Eye Care Insititute, Louisville, Kentucky
  - Central Maine Eye Care, Lewiston, Maine
  - Andover Eye Associates, Andover, Massachusetts
  - Vita Eye Clinic, Shelby, North Carolina
  - Total Eye Care, PA, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SkQ1 Vehicle: Vehicle for SkQ1 ophthalmic solution
Period: Overall Study
Arm/Group | SkQ1 Vehicle | Low Dose - SkQ1 | High Dose - SkQ1
Started | 151 | 150 | 151
Completed | 147 | 144 | 147
Not Completed | 4 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SkQ1 Vehicle | Low Dose - SkQ1 | High Dose - SkQ1 | Total
Number analyzed (Participants) | 151 | 149 | 151 | 451
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 68 | 74 | 87 | 229
  >=65 years | 83 | 75 | 64 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (12.98) | 64.4 (12.35) | 61.4 (13.58) | 63.4 (13.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 99 | 102 | 316
  Male | 36 | 50 | 49 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 14 | 27
  Not Hispanic or Latino | 145 | 142 | 137 | 424
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 2 | 4 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 23 | 14 | 24 | 61
  White | 124 | 130 | 120 | 374
  More than one race | 1 | 1 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 151 | 149 | 151 | 451
Central CFS [Mean (Standard Deviation); unit: units on a scale] | 1.72 (0.73) | 1.67 (0.69) | 1.67 (0.68) | 1.69 (0.70)

OUTCOME MEASURES:

1. Primary Outcome: Central Corneal Staining Change From Baseline
Description: Change of Corneal Fluorescein Staining from baseline to Day 57, scale ranges from 0 to 4, where grade 0 = None, 4 = Severe
Time Frame: From baseline to Day 57
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SkQ1 Vehicle | Low Dose - SkQ1 | High Dose - SkQ1
Number analyzed (Participants) | 151 | 149 | 151
score on a scale | -0.28 (0.773) | -0.3 (0.816) | -0.2 (0.763)

2. Primary Outcome: Grittiness Change From Baseline
Description: Change of patient-reported grittiness from baseline to Day 57, scale ranges from 0 to 5 for each symptom, where 0 = None and 5 = Worst
Time Frame: From baseline to Day 57
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SkQ1 Vehicle | Low Dose - SkQ1 | High Dose - SkQ1
Number analyzed (Participants) | 151 | 149 | 151
score on a scale | -0.42 (1.108) | -0.36 (1.176) | -0.43 (1.387)

ADVERSE EVENTS:
Time Frame: From Day -7 through end of study (Day 57)
Arm/Group | SkQ1 Vehicle | Low Dose - SkQ1 | High Dose - SkQ1
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/149 | 0/151
Serious Adverse Events (participants affected / at risk) | 1/151 | 3/149 | 2/151
Other Adverse Events (participants affected / at risk) | 3/151 | 4/149 | 3/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SkQ1 Vehicle (N=151) | Low Dose - SkQ1 (N=149) | High Dose - SkQ1 (N=151)
Ovarian cancer (Reproductive system and breast disorders) | 0 | 1 | 0
Peripheral arterial occlusive disorder (Vascular disorders) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Procedural pain (Surgical and medical procedures) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SkQ1 Vehicle (N=151) | Low Dose - SkQ1 (N=149) | High Dose - SkQ1 (N=151)
Instillation site pain (General disorders) | 2 | 4 | 3
Visual acuity reduced (Eye disorders) | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship and manuscript composition will reflect cooperation among all parties involved in the study. Authorship will be established before writing the manuscript. The study sponsor will have the final decision regarding the manuscript and publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT03764735/Prot_SAP_000.pdf